CLINICAL TRIAL: NCT03252288
Title: mHealth-Assisted Conditional Cash Transfers to Improve Timeliness of Childhood Vaccinations
Brief Title: mHealth-Assisted Conditional Cash Transfers to Improve Timeliness of Vaccinations (D0271)
Acronym: MINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of South Carolina (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-0591; 1R21TW010262 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Immunization

STUDY DESIGN:
Intervention Model Description: A random event (scheduled vaccination date for a child based on date of birth) will determine whether a women does not receive an intervention (before a certain calendar date) or receives an intervention (after a certain calendar date).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (No Intervention): No intervention
- Reminders only (Experimental): Reminders are sent 1 week and 1 day before each scheduled vaccination date
  Interventions: Behavioral: Reminders
- Reminders + Conditional financial transfer (Experimental): Reminders are sent 1 week and 1 day before each scheduled vaccination date; and conditional financial transfers are made for each on-time vaccination visit
  Interventions: Behavioral: Reminders; Behavioral: Conditional financial transfers

INTERVENTIONS:
Behavioral: Reminders — Text of phone-call based reminders to mobile phones
  Arms: Reminders + Conditional financial transfer; Reminders only
Behavioral: Conditional financial transfers — Full amount paid if visit occurs within 1 week of the scheduled visit; partial amount is paid if visit occurs >1 week but within 4 weeks of the scheduled visit
  Arms: Reminders + Conditional financial transfer

SUMMARY:
Vaccination is a cost-effective strategy for conferring immunity against a host of preventable diseases, however, rates of timely childhood vaccinations remain inadequate in resource-limited settings. We propose to evaluate the feasibility and efficacy of mHealth-assisted conditional cash transfers as a means of overcoming individual barriers to timely vaccinations. The study will form the basis for a pragmatic randomized controlled trial of the efficacy and cost-effectiveness of mHealth reminders and conditional cash transfers for improving rates of timely vaccinations among young children.

DETAILED DESCRIPTION:
Vaccination is one of the most cost-effective strategies for conferring immunity against a host of preventable diseases. The World Health Organization estimates that over 2.5 million child deaths are prevented annually worldwide due to vaccination efforts. Infants must receive all recommended vaccinations in a timely manner to be fully protected from deadly infectious diseases such as tuberculosis, diphtheria, pertussis and polio. A large body of evidence has shown that children living in socio-economically disadvantaged backgrounds are more likely to be vaccinated late, or not at all, compared to their counterparts from wealthier and more educated families. While Tanzania has successfully achieved high national vaccination coverage, there remain substantial regional variations. In this proposal we seek to evaluate the feasibility of combining two emerging types of interventions - mHealth and conditional cash transfers - to overcome individual barriers to timely vaccinations. Researchers at Duke University and Tanzania's National Institute of Medical Research (NIMR) will collaborate to evaluate whether mobile phone (mHealth)-based vaccination reminders, combined with a financial incentive scheme for families with young children, may result in improved vaccination coverage and timeliness. The specific aims of the proposal are to (1) conduct formative research to identify locally relevant client-side and provider-side barriers to timely vaccinations; (2) develop an mHealth system to facilitate and monitor timely vaccinations and conduct surveys with late-stage pregnant women to derive willingness-to-accept estimates and a feasible incentive structure; and (3) assess the efficacy of a combination intervention consisting of mHealth reminders and conditional cash transfers for improving the rates and timeliness of vaccinations among infants in their first 6 months of life. Qualitative follow-up surveys with providers and a subset of clients will assess barriers to the acceptability and scalability of an mHealth supported conditional cash-transfer intervention for timely vaccination. The study will be implemented with support from Tanzania's Ministry of Health and Social Welfare Immunization and Vaccine Development Programme. The results of the proposed study will form the basis for a pragmatic randomized controlled trial of the efficacy and incremental cost-effectiveness of mHealth reminders and conditional cash transfers as means of improving timely vaccinations of young children.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, last trimester
* Access to mobile phone

Exclusion Criteria:

* Cognitive impairment
* Unwillingness to receive study-related information and reminders via mobile phone

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ostermann, MD, PhD, Principal Investigator — University of South Carolina
Locations (1):
- National Institute for Medical Research, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No
Data from the proposed study will be stored in a data repository; this data will be de-identified so that they cannot be linked back to individuals. Investigators wishing to use study data to answer new research questions may submit data analysis concept proposals for consideration by the Principal Investigators. The Principal Investigators will review the proposal and will provide those submitting scientifically rigorous and promising proposals access to the data repository to address their research questions. This will ensure that the data resources of the proposed study will provide the greatest possible benefit to the scientific community.

REFERENCES:
- [Derived] Ostermann J, Hair NL, Moses S, Ngadaya E, Godfrey Mfinanga S, Brown DS, Noel Baumgartner J, Vasudevan L. Is the intention to vaccinate enough? Systematic variation in the value of timely vaccinations and preferences for monetary vs non-monetary incentives among pregnant women in southern Tanzania. Vaccine X. 2023 Jan 23;13:100266. doi: 10.1016/j.jvacx.2023.100266. eCollection 2023 Apr. PMID 36814594
- [Derived] Ostermann J, Vasudevan L, Baumgartner JN, Ngadaya E, Mfinanga SG. Do mobile phone-based reminders and conditional financial transfers improve the timeliness of childhood vaccinations in Tanzania? Study protocol for a quasi-randomized controlled trial. Trials. 2019 Jul 4;20(1):397. doi: 10.1186/s13063-019-3430-4. PMID 31272487

RESULTS

PARTICIPANT FLOW:
Groups:
- No Intervention: No reminders or incentives
- Reminders Only: Reminders are sent 1 week and 1 day before each scheduled vaccination date
  Reminders: Text containing child name and vaccination due date sent via SMS to designated mobile phones
- Reminders + Conditional Financial Transfer: Reminders are sent 1 week and 1 day before each scheduled vaccination date; and conditional financial transfers are made for each on-time vaccination visit
  Reminders: Text containing child name and vaccination due date sent via SMS to designated mobile phones
  Conditional financial transfers: Full amount paid if visit occurs within 1 week of the scheduled visit; partial amount is paid if visit occurs >1 week but within 4 weeks of the scheduled visit
Period: Overall Study
Arm/Group | No Intervention | Reminders Only | Reminders + Conditional Financial Transfer
Started | 239 | 67 | 106
Completed | 140 | 67 | 106
Not Completed | 99 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Death | 11 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 79 | 0 | 0
Not completed — Loss of baseline data on tablets | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of 412 participants enrolled, 14 were disenrolled due to maternal death (n=1), child death (n=11), or withdrawal (n=2), leaving an initial sample of 398 participants. 79 participants were lost to follow-up. Baseline data were lost (due to tablet failure) for 6 participants. The effective enrollment into the trial was N=313. N=310 had valid data on study outcomes and per-protocol assignment to study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention | Reminders Only | Reminders + Conditional Financial Transfer | Total
Number analyzed (Participants) | 140 | 67 | 106 | 313
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 2 | 1 | 18
  Between 18 and 65 years | 125 | 65 | 105 | 295
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 67 | 106 | 313
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 140 | 67 | 106 | 313
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 140 | 67 | 106 | 313
Age [Mean (Standard Deviation); unit: years] | 26.7 (7.56) | 29.7 (6.57) | 30.3 (6.67) | 28.58 (7.24)

OUTCOME MEASURES:

1. Primary Outcome: Number of Timely Vaccinations Received
Description: Number of vaccinations received within 4 weeks of scheduled vaccination dates. Note: Vaccinations are due at birth and at ages 6, 10, and 14 weeks. Delays in 6 and/or 10 week vaccinations result in corresponding shifts in subsequent vaccination due dates. Timeliness is calculated independently for each vaccination in relation to its scheduled due date: The vaccination is considered timely if it is received within 4 weeks of the scheduled due date, not timely otherwise. Observations beyond 6 months after birth are censored.
Time Frame: Up to 6 months after birth
Population: Participants in follow-up survey without missing data on vaccinations and per-protocol study arm
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention | Reminders Only | Reminders + Conditional Financial Transfer
Number analyzed (Participants) | 139 | 67 | 104
Participants
  Received 0 vaccinations within 28 days of target age | 10 | 5 | 5
  Received 1 vaccination within 28 days of target age | 9 | 6 | 12
  Received 2 vaccinations within 28 days of target age | 12 | 6 | 18
  Received 3 vaccinations within 28 days of target age | 27 | 12 | 19
  Received 4 vaccinations within 28 days of target age | 81 | 38 | 50

2. Secondary Outcome: Number of Vaccinations Received
Description: Number of vaccinations received (range 0-4, for the vaccination due at birth, 6, 10, and 14 weeks) Note: Vaccinations are due at birth and at ages 6, 10, and 14 weeks. Delays in 6 and/or 10 week vaccinations result in corresponding shifts in subsequent vaccination due dates. Thus, some vaccinations may be due after the end of the observation period, which ends 6 months after birth).
Time Frame: Up to 6 months after birth
Measure: Count of Participants; unit: Participants
Arm/Group | No Intervention | Reminders Only | Reminders + Conditional Financial Transfer
Number analyzed (Participants) | 139 | 67 | 104
Participants
  Received 0 vaccinations | 0 | 0 | 0
  Received 1 vaccination | 0 | 0 | 0
  Received 2 vaccinations | 1 | 0 | 0
  Received 3 vaccinations | 11 | 11 | 5
  Received 4 vaccinations | 127 | 56 | 99

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Arm/Group | No Intervention | Reminders Only | Reminders + Conditional Financial Transfer
All-Cause Mortality (participants affected / at risk) | 12/239 | 0/67 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/239 | 0/67 | 0/106
Other Adverse Events (participants affected / at risk) | 0/239 | 0/67 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03252288/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03252288/SAP_001.pdf
  • Informed Consent Form (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03252288/ICF_002.pdf